CLINICAL TRIAL: NCT02310360
Title: Measuring Food-induced Striatal and Extra-striatal Dopamine Release Using (18F)Fallypride Positron Emission Tomography
Brief Title: Striatal and Extra-striatal Dopamine Release in Response to Food in Healthy Humans
Acronym: DA-Fallypride
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S56186
Record Dates: First submitted 2014-11-19; First posted 2014-12-08 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Appetite Regulation
MeSH Terms: interventions — fallypride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Healthy volunteers
  Interventions: Radiation: Fallypride

INTERVENTIONS:
Radiation: Fallypride

SUMMARY:
The purpose of this study is to investigate whether a combination of taste probes and food-related cues can induce dopamine release in striatal and extra-striatal brain regions in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 20 ≤ BMI ≤ 25
* Right handed
* Stable body weight for at least 3 consecutive months at start of study and no history of behavioral, therapeutic or surgical treatment aiming at or leading to weight loss/gain
* Subject understands the study procedures and agrees to participate in the study by giving written informed consent

Exclusion Criteria:

* Medical (current or history):

  * Abdominal/thoracic surgery except appendectomy
  * Gastrointestinal, endocrine (especially diabetes), or neurological diseases
  * Cardiovascular, respiratory, renal or urinary diseases
  * Hypertension
  * Food or drug allergies
  * Head trauma with loss of consciousness
* Psychiatric disorders (current or history):

  * Eating disorders
  * Psychotic disorders
  * Major depressive disorder
  * Somatoform disorder
  * Emotional and/or restraint eating
  * Treatment in the last 6 months with antidepressants (as MAO inhibitors), neuroleptics, sedative hypnotics, psychostimulants, glucocorticoids, appetite suppressants, estrogens, opiate, or dopamine medications. Oral contraception is allowed
* History of cannabis use or any other drug of abuse for at least 12 months prior to the study
* Intolerance of lactose
* Vegetarians
* Smoking and alcohol intake greater than 5 alcoholic units per week (one alcoholic unit = 10 gr ethanol)
* More than moderate exercise (> 30 min, five times per week of walking or equivalent)
* High caffeine intake (> 500 ml coffee daily or equivalent)
* Exposure to a significant amount (> 1mSv) of ionizing radiation in other research studies within the last 12 months
* Claustrophobia or too much uneasiness in limited spaces (in order tolerate confinement during PET scanning procedures)
* Inability or unwillingness to perform all of the study procedures, or if the subject is considered unsuitable in any way by the principal investigator
* Recent participation (< 30 days) or simultaneous participation in another clinical trial
* Any condition that would interfere with Magnetic Resonance Imaging (MRI) or PET studies (e.g., cochlear implant, metal fragments in eyes, cardiac pacemaker, neural stimulator, and metallic body inclusion or other metal implanted in the body which may interfere with MRI scanning)
* Anemia
* Pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy females.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
DA release in both striatal and extra-striatal brain regions | 1 year
  A [18F]Fallypride PET protocol and the linearized simplified reference region model (LSSRM) kinetic model will be used to detect DA release.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Van Oudenhove, MD, PhD, Principal Investigator — University Hospitals Leuven, campus Gasthuisberg
Locations (1):
- University Hospitals Leuven, campus Gasthuisberg, Leuven, Belgium